CLINICAL TRIAL: NCT01407458
Title: The Impact of a Structured Physical Activity Program on Bone Strength and Psycho-Motor Learning of Young Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Eias Kassem, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0043-11-HYMC
Record Dates: First submitted 2011-07-26; First posted 2011-08-02 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: Bone Strength; Bone Density

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Active Comparator): Children doing additional exercises with upper limbs in physical education class
  Interventions: Other: Upper Limb Exercises
- Control Group (Active Comparator): Children doing normal physical education exercises
  Interventions: Other: Normal physical exercises

INTERVENTIONS:
Other: Upper Limb Exercises — Upper limb exercises
  Arms: Experimental Group
Other: Normal physical exercises — Exercises usually done by children in physical education classes
  Arms: Control Group

SUMMARY:
To examine the impact of a structured physical activity program focused on bone strength in elementary school children in the framework of their physical education classes on:

1. Bone strength of children participating in the activity.
2. Physical variables and psycho-motor capabilities: vertical jumping strength, horizontal jumping strength, static balance, dynamic balance and coordination.

ELIGIBILITY:
Inclusion Criteria:

* First and second grade pupils
* Healthy

Exclusion Criteria:

* Medical condition does not permit participation in physical education class

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Bone strength | One year
  Examination of bone strength will be carried out by using a measuring device called Sunlight Omnisense. This device uses SOS (Speed of Sound) to check bone strength and density.
Bone density | One year
  Examination of bone density will be carried out by using a measuring device called Sunlight Omnisense. This device uses SOS (Speed of Sound) to check bone strength and density.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel